Title of the study: Long Term Clinical Evaluation of a Posterior Glass Hybrid System vs.

Composite Resin: a Controlled Clinical MultiCenter Study

NCT number: 02717520

Date: November 7<sup>th</sup>, 2019

**Objective:** To evaluate clinical effectiveness of a glass hybrid restorative material as a long-term restorative material in moderate and large size two-surface restorations versus a nano-hybrid composite resin material.

**Study design:** Split-mouth, randomized, prospective and multicentre study.

### **Methods:**

<u>Study population</u>: Healthy patients in need of two surface restorations in the molar region of the same jaw.

### <u>Inclusion criteria</u>:

- 1. Subject > 18 years.
- 2. Subjects with restorative treatments on vital teeth in posterior molar region.
- 3. Subjects with indication for restorative treatment on vital teeth in posterior molar region.
- 4. Restorations limited to two surfaces with one proximal cavity in occlusion.
- 5. Favourable and stable occlusal relationship between the remaining teeth.
- 6. Subject must be reliable, cooperative, and in the opinion of the Investigator, likely to be compliant with study procedures.
- 7. Subject provides written informed consent signed and dated prior to entering the study.

## Exclusion criteria:

- 1. Subject with full dentures or crowns and bridges in oclussal contact with teeth indicated for restorative treatment.
- 2. Subject has a history of drug abuse, addiction to medication or alcohol abuse within the previous year.
- 3. Pulp exposure.
- 4. Known unavailability of subject for recall visit(s).
- 5. Allergy to any ingredient of a material.
- 6. Severe bruxing.
- 7. Subject has a clinically significant or unstable medical or physiological condition.
- 8. Female subject is pregnant or lactating or intends to become pregnant during the course of the study.
- 9. Subject not willing to participate in the study or not able to understand the content of the study

<u>Intervention</u>: Each patient enrolled in the study received one restoration with a glass hybrid material (EQUIA Forte, GC, Tokyo, Japan) and one with a nano- hybrid composite resin material (Tetric EvoCeram, Ivoclar Vivadent, Schaan, Liechtenstein), according to the manufacturers' instructions.

# **Clinical Evaluation**

<u>Recall Periods</u>: One week after placement of the restoration (baseline), and yearly up to 5 years according to the FDI-2 criteria (Hickel et al. 2007; Recommendations for conducting control clinical studies of dental restorative materials. Clin Oral Invest. 2007; 11:5-33).

## Statistical Analysis Plan

Descriptive statistics were primarily implemented. To test the performance of the restorative materials according to the FDI-2 criteria over the study period, Sign test is going to be used and the level of significance is set at  $\alpha$ =0.05.